CLINICAL TRIAL: NCT05669872
Title: A Prospective Randomized Controlled Trial Evaluating the Safety and Efficacy of Patient Blood Management Program in Patients With Gynecologic Cancer
Brief Title: Patient Blood Mangement (PBM) Using IV Iron in Patients With Gynecologic Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Jeong-Yeol Park, MD, PhD, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2022-1674
Record Dates: First submitted 2022-11-29; First posted 2023-01-03 (Actual); Last update posted 2023-01-05 (Actual); Status verified 2023-01

CONDITIONS: Gynecologic Cancer
Keywords: endometrial cancer; ovarian cancer; cervical cancer; patient blood management; IV iron
MeSH Terms: conditions — Endometrial Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms | interventions — ferric carboxymaltose

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- patient blood management group (Experimental): 1. before surgery (within 2-6 weeks before surgery)
     - 7 ≤ Hb < 12 g/dL : ferric carboxymaltose 1000mg
  2. during surgery
     - In case of hemodynamically unstable, transfusion according to the judgment of the operating surgeon and anesthesiologist
  3. after surgery (POD #1)
     * 7 ≤ Hb < 12 g/dL : ferric carboxymaltose 1000mg
     * Hb <7 g/dL : pRBC 2 packs transfusion
  Interventions: Drug: Ferric Carboxymaltose 50Mg/Ml Inj 20Ml
- conventional management group (Active Comparator): 1. before surgery (within 2-6 weeks before surgery)
     * 8 ≤ Hb < 10 g/dL: pRBC 1 pack transfusion
     * Hb < 8 g/dL: pRBC 2 packs transfusion * Use of oral iron supplements, EPO, in control patients is permitted. (no IV iron supplements)
  2. during surgery
     - In case of hemodynamically unstable, transfusion according to the judgment of the operating surgeon and anesthesiologist
  3. after surgery (POD #1)
     * 8 ≤ Hb < 10 g/dL: pRBC 1 pack transfusion
     * Hb < 8 g/dL: pRBC 2 packs transfusion * Use of oral iron supplements, EPO, in control patients is permitted. (no IV iron supplements)
  Interventions: Drug: RBC

INTERVENTIONS:
Drug: Ferric Carboxymaltose 50Mg/Ml Inj 20Ml — ferric carboxymaltose 1000mg, fixed dose for intervention group
  Arms: patient blood management group
Drug: RBC — pack RBC transfusion
  Arms: conventional management group

SUMMARY:
To demonstrate the safety and effectiveness of a patient blood management program in gynecological cancer patients

DETAILED DESCRIPTION:
To demonstrate the safety and effectiveness of a patient blood management program in gynecological cancer patients undergoing surgery, radiation therapy, and chemotherapy, and to establish a patient blood management program and introduce it as a standard treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 20-80 years
2. Untreated, histologically diagnosed cervical cancer, endometrial cancer, and ovarian cancer (including cases diagnosed by imaging without biopsy in the case of ovarian cancer)
3. Patients with ECOG performance status 0-2
4. Patients with ASA PS 1-2
5. Preoperative Hgb ≥ 7 g/dL
6. Patients who are scheduled for preoperative iron panel test (serum ferritin, iron, TIBC)
7. In case of showing proper organ function WBC ≥ 3,000/mm3 Platelets ≥ 100,000/mm3 Creatinine ≤ 2.0 mg/dL Bilirubin ≤ 1.5 x institutional upper limit normal SGOT, SGPT, and ALP ≤ 3 x institutional upper limit normal
8. Patient who voluntarily signed the informed consent form

Exclusion Criteria:

1. Patient who unable to determine whether or not to consent on their own
2. Patients with serious underlying diseases or complications
3. Women who are pregnant or lactating
4. Patients with concurrent infection
5. Patients who are allergic to existing iron preparations
6. Patients who underwent neoadjuvant chemotherapy or preoperative radiation therapy
7. Patients who have had or received cancer treatment within 5 years, except for non-melanoma skin cancer, cervical intraepithelial tumor, and superficial cancer of the stomach and bladder
8. Patients with iron overload or iron utilization disorders
9. Patients with serum ferritin > 800ng/mL or TSAT > 50% on Iron panel tests

Ages: 20 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 334 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
transfusion rate | within 3 weeks after surgery
  Transfusion rate within 3 weeks after surgery, radiation and chemotherapy treatment

SECONDARY OUTCOMES:
hemoglobin differences | within 3 weeks after surgery
  Comparison of hemoglobin differences between the groups
Frequency of anemia | within 3 weeks after surgery
  Frequency of anemia and blood transfusion before adjuvant therapy between the groups
Frequency and delay period of treatment | within 3 weeks after surgery
  Frequency and delay period of treatment delay due to anemia before adjuvant therapy between the groups
The costs that patients actually pay for treatment (Cost-effectiveness) | within 3 weeks after surgery
  Investigate, evaluate, and compare the costs that patients actually pay for treatment between the two groups.
Quality of life of patients EORTC QLQ-C30 | within 3 weeks after surgery
  used to collect information on patients' quality of life and compare the scores of the two groups.
  Scores are given from 1 to 4 for most questions, and the lower the score, the better the patient's quality of life is evaluated. The average of the total scores is used to compare the two groups.
Adverse events | within 3 weeks after surgery
  ADR (adverse drug reaction) is investigated between the two groups, and the rate of adverse reactions and the rate of moderate adverse reactions in each group are compared.
Quality of life of patients HINT-8 | within 3 weeks after surgery
  HINT-8 used to collect information on patients' quality of life and compare the scores of the two groups.
  Each answer is given to 8 questions, and each answer is scored and assigned from 1 to 4 points, and the averages of the two groups are also compared.

CONTACTS AND LOCATIONS:
Overall Officials: Jeong-Yeol Park, Principal Investigator — Asan Medical Center
Locations (1):
- Department of Obstetrics and Gynecology, University of Ulsan College of Medicine, Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Park JY, Kang OJ, Lee YY, Kim YS. A prospective randomized controlled trial evaluating the safety and efficacy of patient blood management program in patients with gynecologic cancer (KGOG 4011/PBM). Int J Gynecol Cancer. 2023 Jul 3;33(7):1140-1144. doi: 10.1136/ijgc-2023-004403. PMID 37094968